CLINICAL TRIAL: NCT01203592
Title: Efficacy of Albuterol in the Treatment of Congenital Myasthenic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andrew Engel, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-004529
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Congenital Myasthenic Syndrome
Keywords: Congenital myasthenic syndrome; Albuterol; Neuromuscular transmission
MeSH Terms: conditions — Myasthenic Syndromes, Congenital | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albuterol (Experimental): 4 mg twice daily by mouth for adults. The dose for children 6 to 12 years is 2 mg two or three times daily; the dose for children 2 to 6 years is 0.1 mg/kg/day (maximum 2 mg) three times daily.
  Interventions: Drug: Albuterol

INTERVENTIONS:
Drug: Albuterol — 4 mg twice daily by mouth for adults. The dose for children 6 to 12 years is 2 mg two or three times daily; the dose for children 2 to 6 years is 0.1 mg/kg/day (maximum 2 mg) three times daily.
  Other Names: Ventolin

SUMMARY:
The study tests the notion that patients suffering from certain types of congenital myasthenic syndromes are benefitted by the use of Albuterol at doses used in clinical practice.

DETAILED DESCRIPTION:
The aim of the proposal is to evaluate the effects of albuterol, an adrenergic agonist, in the treatment of congenital myasthenic syndromes (CMS). Over the past 2 decades I found that some CMS patients refractory to or worsened by cholinergic agonists, namely those suffering from defects in acetylcholinesterase (AChE) or Dok-7, respond to ephedrine, a medication used for over half-a-century in the treatment of autoimmune myasthenia gravis. After ephedrine became unavailable, I treated the same type of patients with albuterol in doses ranging from 4 mg daily to twice daily for adults; the dose for children 6 to 12 years is 2 mg two or three times daily; the dose for children 2 to 6 years is 0.1 mg/kg/day (maximum 2 mg) three times daily. Evaluation of the effects of the medications are based on the Table shown below.

Name:

Mayo Clinic no:

Date of this report: (dd/mm/yyyy):

Before taking Albuterol ER On Albuterol (date of this report)

* Current daily dose of albuterol:

Dates when started (d/m/year) Daily dose Distance in feet walked without stopping to rest Number of steps climbed without stopping to rest Difficult to sit up from lying on back* Difficult to rise from sitting* Difficult to speak or swallow* Shortness of breath on exertion* Shortness of breath at night* Weakness of arm or hand muscles * Weakness of leg or foot muscles*

*Rate as mild, moderate, severe Describe below any additional changes in your condition such as arm elevation time, number of deep knee bends before having to stop, or in activities of daily living relevant to the effects of the treatment. Also indicate any unwanted side effects of the medication. Continue on other side or separate page if necessary. Return this questionnaire to Dr. Andrew Engel (email:schaefer.cleo@mayo.edu) ,after treatment with albuterol for 1 month and then monthly thereafter, or mail to Dr. Andrew Engel, Department of Neurology, Mayo Clinic, Rochester, MN 55905.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital myasthenic syndrome substantiated by typical clinical history, seronegativity to AChR and MuSK, and evidence of a decremental EMG response.

Exclusion Criteria:

* Uncontrolled hypertension, arrhythmias, or other significant cardiac disease.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Name: Efficacy of albuterol in the treatment of congenital myasthenic syndromes | 3 years
  The primary outcome measures pertain to evaluating the improvement in the patient's strength

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Engel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States